CLINICAL TRIAL: NCT06650761
Title: A Randomized, Double-Blind, Placebo-Controlled, Three-Part, Phase 1a Dose Escalation Clinical Trial to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CDX-622 in Healthy Participants
Brief Title: A Phase I Study of CDX-622
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDX622-01
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CDX-622 (Experimental): Eligible participants will receive doses of CDX-622 by IV or SC
  Interventions: Drug: CDX-622
- Normal Saline (Placebo Comparator): Eligible participants will receive doses of Normal Saline by IV or SC
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: CDX-622 — Up to 4 infusions of one of seven dosages of CDX-622 or up to 1 dose by subcutaneous injection of one of three dosages of CDX-622
  Arms: CDX-622
Drug: Normal Saline — Up to 4 infusions or 6 SC injections of normal saline
  Arms: Normal Saline

SUMMARY:
This is a study to determine the safety of CDX-622 in healthy participants.

DETAILED DESCRIPTION:
CDX-622 is a bispecific antibody that binds to stem cell factor (SCF) and thymic stromal lymphopoietin (TSLP).

This study will evaluate the safety, pharmacokinetics, and Pharmacodynamics of IV single ascending doses (Part 1), IV multiple ascending doses (Part 2), and subcutaneous (SC) single ascending doses (Part 3) of CDX-622 in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* An informed consent signed and dated by the participant.
* Healthy volunteer aged 18-55.
* In generally good health and without significant medical conditions based on physical exam, ECG, and laboratory test results.
* Body mass index (BMI) ≥ 18 kg/m2 to ≤ 32 kg/m2.
* No course of medication, whether prescribed or over the counter, in the 4 weeks before study drug administration.
* Both males and females of childbearing potential must agree to use a medically accepted contraceptive regimen during study and up to 150 days afterwards.
* Not a current smoker (or regular user of any nicotine containing product).
* Willing to follow all study rules.

Key Exclusion Criteria:

* Women who are pregnant or nursing.
* History of anaphylaxis, food allergies, or allergies (chronic or seasonal) requiring prescription medication.
* History of asthma requiring the use of inhaled medication within the past 5 years.
* Vaccination within 4 weeks prior to study drug administration (subjects must agree to avoid vaccination during the study).
* Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to Screening.
* Positive urine test for alcohol and drugs of abuse.

Additional protocol defined inclusion and exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Trials. Infusion reactions will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | Day 1 up to Day 127
  To evaluate the safety profile as determined by the incidence of adverse events in single or multiple ascending doses of CDX-622 or placebo comparator in healthy participants.

SECONDARY OUTCOMES:
CDX-622 serum evaluations over time | Day 1 up to Day 127
  CDX-622 serum concentrations will be measured at specified visits
CDX-622 biomarker evaluations over time | Day 1 up to Day 127
  The effect of CDX-622 on serum tryptase levels and other relevant biomarkers
Measurement of anti-drug antibody development over time | Day 1 up to Day 127
  Participants will be monitored for the development of anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States